CLINICAL TRIAL: NCT06292013
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Effect of Lepodisiran on the Reduction of Major Adverse Cardiovascular Events in Adults With Elevated Lipoprotein(a) Who Have Established Atherosclerotic Cardiovascular Disease or Are at Risk for a First Cardiovascular Event - ACCLAIM-Lp(a)
Brief Title: A Study to Investigate the Effect of Lepodisiran on the Reduction of Major Adverse Cardiovascular Events in Adults With Elevated Lipoprotein(a) - ACCLAIM-Lp(a)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18812; J3L-MC-EZEF (Other: Eli Lilly and Company); 2023-509190-23 (EudraCT Number)
Record Dates: First submitted 2024-02-27; First posted 2024-03-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Elevated Lp(a)
Keywords: ASCVD; LY3819469; lepodisiran
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lepodisiran Sodium (Experimental): Lepodisiran sodium administered subcutaneously (SC).
  Interventions: Drug: Lepodisiran Sodium
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lepodisiran Sodium — Administered SC
  Other Names: LY3819469
  Arms: Lepodisiran Sodium
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of lepodisiran in reducing cardiovascular risk in participants with high lipoprotein(a) who have cardiovascular disease or are at risk of a heart attack or stroke. The study drug will be administered subcutaneously (SC) (under the skin). Approximately 1700 additional participants will be enrolled in an addendum to explore Lp(a) lowering with an alternative dosing schema.

ELIGIBILITY:
Inclusion Criteria:

* Have Lipoprotein(a) [Lp(a)] ≥175 nanomoles per liter (nmol/L).
* Meet criteria of either 2a or 2b:

  2a: Individuals 18 years of age or older with established atherosclerotic cardiovascular disease (ASCVD) with an event or revascularization.

  2b: Individuals 55 years of age or older who are at risk for a first cardiovascular (CV) event and either: Documented coronary artery disease (CAD), carotid stenosis, or peripheral artery disease (PAD) without history of event or revascularization; known familial hypercholesteremia; or a combination of high-risk factors.

Exclusion Criteria:

* Have had a major cardiovascular event or surgery, such as myocardial infarction (MI), stroke or coronary or peripheral revascularization, < 60 days before screening
* Have uncontrolled hypertension
* Have New York Heart Association class IV heart failure.
* Have lipoprotein apheresis within 90 days of screening, or planned lipoprotein apheresis during the study.
* Have severe renal failure, defined as

  * Estimated glomerular rate (eGFR) <15 milliliters per minute per 1.73 meters squared (mL/min/1.73m2) at screening Visit 1, or ongoing dialysis.
* Have a diagnosis of active nephrotic syndrome, or urine albumin-creatinine ratio (UACR) of ≥5000 mg/g at screening Visit 1.
* Have acute or chronic hepatitis, known cirrhosis, signs and symptoms of any other liver disease other than metabolic-associated steatotic liver disease, or exclusionary laboratory results as determined by the central laboratory during screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17300 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Any Component of the Major Adverse Cardiac Event (MACE)-4 Composite Endpoint | Baseline up to End of Study (About 4.5 Years)
  Time to first event in a MACE-4 composite endpoint, comprised of cardiovascular death, nonfatal myocardial infarction, nonfatal ischemic stroke, and urgent coronary revascularization.

SECONDARY OUTCOMES:
Change from Baseline in Lipoprotein(a) [Lp(a)] at Week 4 | Baseline, Week 4
  Change from Baseline in Lp(a)
Time to First Occurrence of Any of the Component of MACE-3 Composite Endpoint | Baseline up to End of Study (About 4.5 Years)
  Time to first occurrence MACE-3
Time to First Occurrence of Fatal or Non-Fatal Myocardial Infarction | Baseline up to End of Study (About 4.5 Years)
  Time to first occurrence of fatal or non-fatal myocardial infarction.
Time to Cardiovascular Death | Baseline up to End of Study (About 4.5 Years)
  Time to cardiovascular death.
Time to Occurrence of All-Cause Death | Baseline up to End of Study (About 4.5 Years)
  Time to occurrence of all-cause death
Time to First Occurrence of Any Component of the MACE-4 Composite Endpoint (In the Population with Established ASCVD and CV Event, or Revascularization) | Baseline up to End of Study (About 4.5 Years)
  Time to first occurrence of any component of the MACE-4 composite endpoint.
Time to First Occurrence of any Component of the MACE-4 Composite Endpoint (In the Population At Risk for First CV event) | Baseline up to End of Study (About 4.5 Years)
  Time to first occurrence of any component of the MACE-4 composite endpoint.
Time to First Occurrence of any Component of the MACE-4 Composite Endpoint (In the Population with Lp(a) ≥ 200 nmol/L) | Baseline up to End of Study (About 4.5 Years)
  Time to first occurrence of any component of the MACE-4 composite endpoint.
Time to First Occurrence of Any Component of MACE-3 + MALE Composite Endpoint | Baseline up to End of Study (About 4.5 Years)
  Time to first occurrence of any component of MACE-3 + MALE composite endpoint.
Time to First Occurrence of Any Component of Coronary MACE-3 Composite Endpoint | Baseline up to End of Study (About 4.5 Years)
  Time to first Occurrence of any component of coronary MACE-3 composite endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (928):
- United States (222):
  - Birmingham Clinical Research, Birmingham, Alabama
  - Alliance for Multispecialty Research, LLC, Daphne, Alabama
  - SEC Clinical Research, Dothan, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Mobile Heart Specialists, Mobile, Alabama
  - Prime Medical Group, LLC dba Gilbert Center for Family Medicine, LLC, Gilbert, Arizona
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Sun City Clinical Research, Glendale, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Helios Clinical Research - Phoenix, Phoenix, Arizona
  - Absolute Clinical Research, Phoenix, Arizona
  - Clinical Research Institute of Arizona (CRI) - Sun City West, Sun City West, Arizona
  - Pima Heart, Tucson, Arizona
  - Synexus Clinical Research US, Inc./Orange Grove Family Practice, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - National Heart Institute, Beverly Hills, California
  - Valley Clinical Trials, Inc., Covina, California
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - HB Clinical Trials - Fountain Valley, Fountain Valley, California
  - Care Access - Huntington Beach, Huntington Beach, California
  - 310 Clinical Research, Inglewood, California
  - UCSD - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - First Valley Medical Group, Lancaster, California
  - MemorialCare Health System - Long Beach Medical Center, Long Beach, California
  - Ark Clinical Research, Long Beach, California
  - Keck School of Medicine of USC, Los Angeles, California
  - Cardiovascular Research Foundation of Southern California, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Care Access - Santa Clarita, Santa Clarita, California
  - Stanford University Medical Center, Stanford, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Care Access - Thousand Oaks, Thousand Oaks, California
  - Med Partners, Inc. dba Premiere Medical Center of Burbank, Inc., Toluca Lake, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - UCLA South Bay Endocrinology, Torrance, California
  - InvivoCure, Van Nuys, California
  - Synexus Clinical Research US, Inc., Vista, California
  - Interventional Cardiology Medical Group, West Hills, California
  - Millennium Clinical Trials, Westlake Village, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Hartford Hospital (HH), Hartford, Connecticut
  - Cardiology Associates of Fairfield County, P.C., Stamford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Clearwater Cardiovascular & Interventional Consultants M.D., P.A., Clearwater, Florida
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Jellinger and Lerman, MD PA dba The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Elite Cardiac Research Center, Hialeah, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clearwater Cardiovascular & Interventional Consultants M.D., P.A., Largo, Florida
  - K2 Medical Research - Maitland, Maitland, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Flourish Research - Miami, LLC, Miami, Florida
  - Inpatient Research Clinic, Miami Lakes, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida
  - Renstar Medical Research, Ocala, Florida
  - CTR Oakwater, LLC, Orlando, Florida
  - Florida Institute For Clinical Research, LLC, Orlando, Florida
  - Innovative Research Institute - Port Charlotte, Port Charlotte, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clearwater Cardiovascular & Interventional Consultants M.D., P.A., Safety Harbor, Florida
  - Care Access - Tamarac, Tamarac, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Care Access - Tampa, Tampa, Florida
  - Cardiology Partners Clinical Research Institute - Wellington, Wellington, Florida
  - American Clinical Trials - Acworth, Acworth, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Southeastern Clinical Research Institute, Augusta, Georgia
  - East Coast Institute for Research - Canton, Canton, Georgia
  - American Clinical Trials - Douglasville, Douglasville, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Georgia Clinical Research - Lawrenceville, Lawrenceville, Georgia
  - The Jones Center Clinical Research, Macon, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - CARE Institute, Meridian, Idaho
  - Chicago Clinical Research Institute, Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Clinical Investigation Specialists, Gurnee, Illinois
  - Alliance for Multispecialty Research, LLC, Park Ridge, Illinois
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - Accellacare - DuPage, Winfield, Illinois
  - American Health Network of Indiana, LLC - Avon, Avon, Indiana
  - American Health Network of Indiana, LLC - Franklin, Franklin, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Care Access - South Indianapolis, Indianapolis, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Qualmedica Research, Bowling Green, Kentucky
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Grace Research - Bossier, Bossier City, Louisiana
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - IMA Clinical Research, Monroe, Louisiana
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Louisiana Heart Center - Slidell, Slidell, Louisiana
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Care Access - Baltimore, Baltimore, Maryland
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Jadestone Clinical Research, Beltsville, Maryland
  - Flourish Research - Bowie, Bowie, Maryland
  - Kur Research - Columbia Medical, Columbia, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - Brigham and Women's Hospital Diabetes Program, Boston, Massachusetts
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Care Access - Quincy, Quincy, Massachusetts
  - Alliance for Multispecialty Research, LLC., Dearborn, Michigan
  - Revival Research Institute, LLC, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Michigan Heart & Vascular Institute, Ypsilanti, Michigan
  - The National Diabetes & Obesity Research Institute, Diamondhead, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Las Vegas Endocrinology, Henderson, Nevada
  - DaVita Clinical Research - Las Vegas, Las Vegas, Nevada
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - Internal Medicine Associates, Bridgeton, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - Atlantic Health System Overlook Medical Center, Summit, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - IMA Clinical Research, Albuquerque, New Mexico
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - St. Francis Hospital & Heart Center, New Hyde Park, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - IMA Clinical Research Manhattan, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Northwell Health Physician Peconic, Riverhead, New York
  - University of Rochester Medical Center, Rochester, New York
  - Saratoga Clinical Research, Saratoga Springs, New York
  - Stony Brook University, Stony Brook, New York
  - Care Access - Fayetteville, Fayetteville, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Physician's East Endocrinology, Greenville, North Carolina
  - IMA Clinical Research Mount Airy, Mount Airy, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Velocity Clinical Research, Cleveland, Beachwood, Ohio
  - Velocity Clinical Research, Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research, Springdale, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Good Samaritan Regional Medical Center, Corvallis, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Heritage Valley Multispecialty Group, Inc, Beaver, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Abington Medical Specialists, Horsham, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Keystone Clinical Studies, Plymouth Meeting, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Cardiology Consultants of Philadelphia Yardley, Yardley, Pennsylvania
  - Heart and Vascular Research at WellSpan Health, York, Pennsylvania
  - Accellacare Trident Cardiology, Charleston, South Carolina
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Walker Family Care, Little River, South Carolina
  - Care Access - Mauldin, Mauldin, South Carolina
  - Accellacare - Mt Pleasant, Mt. Pleasant, South Carolina
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Care Access - Memphis 2, Memphis, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - Amarillo Heart Clinical Research Institute Inc., Amarillo, Texas
  - IMA Clinical Research Austin, Austin, Texas
  - Velocity Clinical Research, Austin, Austin, Texas
  - Headlands Horizons LLC, Brownsville, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - Private Practice - Dr. James E. Race, Dallas, Texas
  - Baylor Soltero CV Research Center, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Cardio Voyage, Denison, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Texas Health Research & Education Institute - Fort Worth, Fort Worth, Texas
  - Center for Cardiometabolic Disease Prevention/Baylor College of Medicine, Houston, Texas
  - Juno Research, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Accurate Clinical Research - Humble, Humble, Texas
  - The Heart Institute of East Texas, Lufkin, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Wellness Clinical Research, McKinney, Texas
  - North Texas Research Associates, McKinney, Texas
  - Revival Research Institute, LLC, McKinney, Texas
  - Texas Institute of Cardiology, PA, McKinney, Texas
  - PRX Research, Mesquite, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - DaVita Clinical Research - North Houston, Shenandoah, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Alpine Research Organization, Clinton, Utah
  - Intermountain Medical Center, Murray, Utah
  - Virginia Heart, Falls Church, Virginia
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia
  - Eastside Research Associates, Redmond, Washington
  - IMA Clinical Research West Virginia, Morgantown, West Virginia
  - Clinical Investigation Specialists, Kenosha, Wisconsin
- Argentina (54):
  - Clínica Privada del Prado SRL, Alberdi
  - Buenos Aires Macula S.A, Buenos Aires
  - Instituto Médico Especializado (IME), Buenos Aires
  - Consultorio Medico Dr Litvak Bruno, Buenos Aires
  - Consultorio Medico Investigador Principal Dr Besada, Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - CIPREC, Buenos Aires
  - Fundación favaloro para la Docencia e Investigación Médica, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Centro Médico Arsema, Buenos Aires
  - Glenny Corp. S.A., Buenos Aires
  - CEDIC, CABA
  - IDIM - Instituto de Investigaciones Metabólicas, Ciudad de Buenos Aires
  - Instituto de Cardiología "Juana F. Cabral", Corrientes
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Sanatorio Privado Duarte Quirós, Córdoba
  - Centro Médico Colón, Córdoba
  - CIDIM-Centro Integral de Diagnostico por Imagenes Marchegiani, Córdoba
  - MICA - Medicina e Investigación Cardiometabólica, Del Viso
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Hospital Italiano de La Plata, La Plata
  - CIMeL, Lanús
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - Instituto de Cardiología Wolff, Mendoza
  - Clínica Privada Independencia, Munro
  - Centro Privado de Medicina Respiratoria, Paraná
  - CER medical Institute, Quilmes
  - Instituto De Investigaciones Clinicas Quilmes, Quilmes
  - DIM Clínica Privada, Ramos Mejía
  - Instituto Médico Río Cuarto, Río Cuarto
  - Fundacion Estudios Clinicos, Rosario
  - INECO Neurociencias Oroño, Rosario
  - Instituto Especialidades de la Salud Rosario, Rosario
  - Instituto Médico Catamarca IMEC, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Laboratorio de Hemostasia y Trombosis, Rosario
  - Hospital Provincial del Centenario, Rosario
  - Centro Cardiovascular Salta, Salta
  - Corporación Médica San Martín, San Martín
  - Centro Modelo de Cardiología, San Miguel de Tucumán
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán
  - Go Centro Medico San Nicolás, San Nicolás
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares, Santa Fe
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Sanatorio San Martin, Venado Tuerto
- Australia (32):
  - Nightingale Research, Adelaide
  - Advara HeartCare Leabrook, Adelaide
  - Paratus Clinical Research Western Sydney, Blacktown
  - Emeritus Research, Botany
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Core Research Group, Brisbane
  - Heart of Australia, Brisbane
  - Cholesterol Care, Brisbane
  - Paratus Clinical Research Canberra, Bruce
  - Emeritus Research, Camberwell
  - Victorian Heart Hospital, Clayton
  - Barwon Health, Geelong
  - Austin Health - Repatriation Hospital, Heidelberg West
  - Paratus Clinical Research Brisbane, Herston
  - Advara HeartCare Joondalup, Joondalup
  - Paratus Clinical Research Central Coast, Kanwal
  - Liverpool Hospital, Liverpool
  - Logan Hospital, Meadowbrook
  - University of the Sunshine Coast (UniSC) Clinical Trials - Meadowbrook, Meadowbrook
  - AusTrials - Sunshine, Melbourne
  - The AIM Centre / Hunter Diabetes Centre, Merewether
  - USC Clinical Trials Moreton Bay, Morayfield
  - Advara HeartCare - Mulgrave, Mulgrave
  - University of the Sunshine Coast (UniSC) Clinical Trials - Noosa, Noosaville
  - Fusion Clinical Research, Norwood
  - Clinitrials, Perth
  - Royal Perth Hospital, Perth
  - USC Clinical Trials Sunshine Coast, Sippy Downs
  - USC Clinical Trials Brisbane (South Bank), South Brisbane
  - Momentum St. Leonards, Sydney
  - Townsville University Hospital, Townsville
- Austria (15):
  - Krankenhaus St. Josef Braunau, Braunau am Inn
  - VIVIT, Feldkirch
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Konventhospital der Barmherzigen Brüder Linz, Linz
  - Landesklinikum Mistelbach, Mistelbach
  - Uniklinikum Salzburg, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Klinik Landstraße, Vienna
  - Zentrum für klinische Studien Dr Hanusch Gmbh, Vienna
  - Medizinische Universität Wien, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
  - Herz Zentrum Währing - Innere Medizin und Kardiologie | Alle Kassen und Privat, Vienna
  - Klinik Floridsdorf, Vienna
- Belgium (18):
  - ZAS Middelheim, Antwerp
  - Imelda General Hospital, Bonheiden
  - Algemeen Ziekenhuis klina, Brasschaat
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - AZ Sint-Blasius, Dendermonde
  - Antwerp University Hospital, Edegem
  - Ziekenhuis Oost-Limburg, Campus St.-Jan, Genk
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - AZ Sint-Maarten, Mechelen
  - AZ Oostende vzw, Ostend
  - AZ Delta vzw, Roeselare
- Brazil (50):
  - Centro de Pesquisa Clinica do Coracao, Aracaju
  - Instituto Aramari Apo, Asa Norte
  - Hospital Universitário João de Barros Barreto, Belém
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Freire Pesquisa Clínica, Belo Horizonte
  - NUPEC - Cardio, Belo Horizonte
  - AngioKormann Blumenau, Blumenau
  - L2IP - Instituto de Pesquisas Clínicas, Brasília
  - Instituto D'Or de Pesquisa e Ensino (IDOR) - Filial Brasília, Brasília
  - Chronos Pesquisa Clínica, Brasília
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Sao Lucas, Campinas
  - Quanta Diagnóstico e Terapia, Curitiba
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR, Curitiba
  - Nucleo De Pesquisa Clinica, Curitiba
  - Universidade Federal de Goias, Goiânia
  - Centro de Pesquisas Clínicas Dr. Marco Mota, Maceió
  - Instituto Do Coracao De Marilia, Marília
  - CHN - Complexo Hospitalar de Niterói, Niterói
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital Moinhos de Vento, Porto Alegre
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Hospital Nossa Senhora da Conceição, Porto Alegre
  - CAPED Centro Avancado Pesquisa e Diagnostica, Ribeirão Preto
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Instituto D'Or Pesquisa e Ensino, Rio de Janeiro
  - Instituto D'Or de Pesquisa e Ensino (IDOR) - Filial Salvador, Salvador
  - Hospital Ana Nery (HAN) - Salvador, Salvador
  - Hospital Da Bahia, Salvador
  - Faculdade de Medicina do ABC, Santo André
  - Praxis Pesquisa Medica, Santo André
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - Centro Internacional de Pesquisa Clínica (CIPES), São José dos Campos
  - CPQuali Pesquisa Clínica, São Paulo
  - CPCLIN, São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital do Coracao, São Paulo
  - Instituto Dante Pazzanese de Cardiology, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Incor - Instituto do Coracao, São Paulo
  - Instituto de Molestias Cardiovasculares de Tatui, Tatuí
  - Eurolatino Pesquisas Medicas, Uberlândia
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Canada (27):
  - Cardio Health Clinical Trial - Brampton, Brampton
  - Ecogene-21, Chicoutimi
  - Viacar Recherche Clinique, Greenfield Park
  - Premier Clinical Trial Network, Hamilton
  - Diex Recherche Inc. Division Joliette, Joliette
  - Milestone Research Inc., London
  - Cardio Health Clinical Trial - London, London
  - G A Research Associates, Moncton
  - Fraser Clinical Trials Inc, New Westminster
  - The Medical Arts Health Research Group, North Vancouver
  - North York Diagnostic and Cardiac Centre, North York
  - Oakville Cardiovascular Research LP, Oakville
  - Medical Arts Health Research Group, Penticton
  - Clinique des Maladies Lipidiques de Québec, Québec
  - ALPHA Recherche Clinique, Québec
  - Unité de Recherche Clinique du CISSS des Laurentides, Saint-Jérôme
  - Cardio Health Clinical Trial - St. Thomas, St. Thomas
  - SMH Cardiology Clinical Trials, Surrey
  - Care Access - Cape Breton, Sydney
  - Centre de Medecine Metabolique de Lanaudiere (CMML), Terrebonne
  - Corcare, Toronto
  - Diabetes Heart Research Centre, Toronto
  - Diex Recherche Inc. Division Trois-Rivieres, Trois-Rivières
  - ARC Biosystems, Vancouver
  - Victoria Heart Institute Foundation, Victoria
  - Discovery Clinical Services, Victoria
  - Winnipeg Clinic, Winnipeg
- China (62):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - China-Japan Union Hospital, Changchun
  - Changde First People's Hospital, Changde
  - The Third Xiangya Hospital of Central South University, Changsha
  - Changzhou Second People's Hospital, Changzhou
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Chifeng Hospital, Chifeng
  - 2nd Affiliated Hospital Chongqing Medical Universi, Chongqing
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian
  - Shunde Hospital of Southern Medical Univesity, Foshan
  - Guangdong Provincial People's Hospital, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Hospital of Harbin Medical University, Harbin
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The Second People's Hospital of Hefei, Hefei
  - Inner Mongolia People's Hospital, Hohhot
  - Huizhou Municipal Central Hospital, Huizhou
  - Jinan Central Hospital, Jinan
  - Jingzhou Central Hospital, Jingzhou
  - The First Hospital of Lanzhou University, Lanzhou
  - Lishui Central Hospital, Lishui
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The Third Hospital of Nanchang, Nanchang
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Guangxi People's Hospital, Nanning
  - Nanyang Second General Hospital, Nanyang
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - Ningbo First Hospital, Ningbo
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital,Fudan University, Shanghai
  - Shanghai Putuo District Center Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shanghai No. 6 People's Hospital - Jinshan Central Hospital, Shanghai
  - The People's Hospital of Liaoning Province, Shenyang
  - Shenzhen Sun Yat-sen Cardiovascular Hospital, Shenzhen
  - Siping Central People's Hospital, Siping
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Fourth Centre Hospital, Tianjin
  - TEDA International Cardiovascular Hospital, Tianjin
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Chongqing Three Gorges Central Hospital, Wanzhou
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan University Medical College - Hubei Zhongshan Hospital, Wuhan
  - Wuhan Asia Heart Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Tangdu Hospital of Fourth Military Medical University of Chinese People's Liberation Army, Xi'an
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Shaanxi provincial people's hospital, Xi'an
  - Xiamen Cardiovascular Hospital, Xiamen
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - General Hospital of Ningxia Medical University, Yinchuan
  - The First People's Hospital of Yueyang, Yueyang
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zigong First People's Hospital, Zigong
- Czechia (21):
  - MEDICUS SERVICES s.r.o., kardiologicka ambulance, Brandýs nad Labem-Stará Boleslav
  - Fakultni Nemocnice u sv. Anny v Brne, Brno
  - Kardiologická ambulance Brno, Brno
  - EFERTUS healthcare s.r.o., Brno
  - Vojenská Nemocnice Brno, Brno
  - Kardiologicka ambulance, Litovel
  - EDUMED - Náchod, Náchod
  - Agentura Science Pro, Olomouc
  - PreventaMed, Olomouc
  - Kardiologicka a Angiologicka Ambulance, Ostrava
  - Private Practice - Dr. Miroslav Koliba, Ostrava
  - Kardio Uhrineves, Prague
  - Synexus Czech, Prague
  - Angiocentrum Komorany, Prague
  - Nefrologie, Prague
  - Poliklinika Lípa Centrum, Prague
  - Centrum Kardiovaskularni Mediciny, Prague
  - Nova kardiologie - Kardiologicka ambulance, Říčany
  - Kardiologicka ambulance MUDr. Ferkl s.r.o., Trutnov
  - Clinical Trials Service s.r.o., Uherské Hradiště
  - Cardio Research, s.r.o, Zlín
- Denmark (9):
  - Sygehus Sønderjylland i Aabenraa, Aabenraa
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Rigshospitalet, Copenhagen
  - Esbjerg sygehus, Syddansk Universitetshospital, Esbjerg
  - Sanos Clinic - Nordjylland, Gandrup
  - Herlev and Gentofte Hospital, Herlev
  - Sanos Clinic, Herlev
  - Holbæk Sygehus, Holbæk
  - Sanos Clinic - Syddanmark, Vejle
- France (25):
  - Hôpital Avicenne, Bobigny
  - Hospices Civils de Lyon - Hopital Louis Pradel, Bron
  - CHRU Troussau, Chambray-lès-Tours
  - Centre Hospitalier Compiègne-Noyon, Compiègne
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Hopital Claude Huriez - CHU de Lille, Lille
  - Centre Hospitalier Saint Joseph - Saint Luc, Lyon
  - Hôpital de la Conception, Marseille
  - Hôpital Saint Joseph, Marseille
  - CHU Montpellier Lapeyronie Hospital, Montpellier
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Centre Hospitalier Universitaire de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Pitie Salpetriere University Hospital, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat - Claude-Bernard, Paris
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier de Pau, Pau
  - CHU Bordeaux Haut-Leveque, Pessac
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes
  - CHU Charles Nicolle, Rouen
  - CHU Strasbourg-Hautepierre, Strasbourg
  - CHU Rangueil, Toulouse
  - Polyclinique Vauban, Valenciennes
- Germany (32):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum am Plattenwald, Bad Friedrichshall
  - Zentrum für klinische Studien Bad Homburg, Bad Homburg
  - Kardiologische Praxen im Spreebogen, Berlin
  - Praxis Rankestrasse, Berlin
  - DRK Kliniken Berlin - Köpenick, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Klinikum Bielefeld Mitte, Bielefeld
  - Universitaetsklinikum Koeln, Cologne
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller GmbH/Zentrum für klinische Studien, Dresden
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Medizentrum Essen Borbeck, Essen
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - BAG Diabeteszentrum Dr. Tews & Partner, Gelnhausen
  - Cardiologicum Hamburg, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Herzzentrum Leipzig GmbH, Leipzig
  - Praxis Oedeme, Lüneburg
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - ze:ro ARZTPRAXEN, Mannheim
  - Universitätsmedizin Mannheim, Mannheim
  - Deutsches Herzzentrum München, Munich
  - Institut für Diabetesforschung GmbH Münster, Münster
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam
  - Universitätsklinikum Regensburg, Regensburg
  - Universitaet zu Koeln - Sana-Klinikum Remscheid GmbH - Klinik fuer Kardiologie, Pneumologie und Internisti -T, Remscheid
  - GPR Gesundheits- und Pflegezentrum Rüsselsheim, Rüsselsheim am Main
  - Zentrum für klinische Studien, Saint Ingbert
  - Studienzentrum Herzklinik Ulm MVZ, Ulm
- Greece (9):
  - Athens Naval Hospital, Athens
  - General Hospital of Athens Laiko, Athens
  - Athens Medical Center, Athens
  - Attikon General University Hospital, Chaïdári
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - Iatriko Paleou Falirou Medical Center, Palaió Fáliro
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Hungary (8):
  - DRC Gyógyszervizsgáló Központ, Balatongyörök
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - Semmelweis University, Budapest
  - Privát Doktor Egészségügyi Zrt, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Medifarma 98 Kft, Nyíregyháza
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Vita Verum Medical Egeszsegugyi Szolgaltato, Székesfehérvár
- India (10):
  - KLES Dr. Prabhakar Kore Hospital & M.R.C, Belagavi
  - Sardar Patel Medical College, Bikaner
  - Shri Mahant Indiresh Hospital, Dehradun
  - K care Hospital, Kanpur
  - Lisie Hospital, Kochi
  - Government Medical College - Kozhikode, Kozhikode
  - King George's Medical University, Lucknow
  - Vijan Hospital & Research Centre, Nashik
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - All India Institute of Medical Sciences, Raipur
- Israel (15):
  - Emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Carmel Hospital, Haifa
  - Linn Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Clalit Health Services - Sakhnin Community Clinic, Sakhnin
  - Sourasky Medical Center, Tel Aviv
- Italy (14):
  - Ospedale Cazzavillan di Arzignano, Arzignano
  - Ospedale di Baggiovara, Baggiovara
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Ospedale Bassini, Cinisello Balsamo
  - Azienda Ospedaliero Universitaria S.Anna, Ferrara
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Martino, Genova
  - Centro Cardiologico Monzino, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedale - Università Padova, Padua
  - Hospital Santa Maria della Misericordia in Perugia, Perugia
  - Fondazione G. Monasterio, Pisa
  - AOU Policlinico Umberto I, Rome
- Japan (68):
  - Asahi Hospital - Asahi, Asahi
  - Asahikawa City Hospital, Asahikawa
  - Saiseikai Futsukaichi Hospital, Chikushino-shi
  - University of Yamanashi Hospital, Chūō
  - The Institute of Medical Science, Asahi Life Foundation, Chūōku
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Fukuwa Clinic, Chūōku
  - Fukuoka Wajiro Hospital, Fukuoka
  - Hakodate Municipal Hospital, Hakodate
  - Public Matto Ishikawa Central Hospital, Hakusan
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji
  - Tokai University Hospital, Isehara
  - Rinku General Medical Center, Izumisano
  - Tenyoukai Central Clinic, Kagoshima
  - Takai Internal Medicine Clinic, Kamakura-shi
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - Kanazawa University Hospital, Kanazawa
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Kasugai Municipal Hospital, Kasugai
  - Kokura Memorial Hospital, Kitakyushu
  - Kobe City Medical Center General Hospital, Kobe
  - Komatsu Municipal Hospital, Komatsu
  - Jinnouchi Hospital, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - Chugoku Rosai Hospital, Kure
  - Rakuwakai Marutamachi Hospital, Kyoto
  - Rakuwakai Otowa Hospital, Kyoto
  - Aizawa Hospital, Matsumoto
  - National Hospital Organization Tokyo Medical Center, Meguro-ku
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Miyakonojo Medical Association Hospital - Tarobocho, Miyakonojō
  - Miyazaki Medical Association Hospital, Miyazaki
  - Iwate Prefectural Central Hospital, Morioka
  - Kanazawa Medical University Hospital, Mukai-awagasaki
  - Tachikawa Medical Center, Nagaoka
  - Nagoya City University Hospital, Nagoya
  - Shonan Oiso Hospital, Naka-gun
  - Nogata Clinic, Nakano
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - National Hospital Organization Okayama Medical Center, Okayama
  - Medical Corporation Sato Medical clinic, Ootaku
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research, Osaka
  - Osaka Keisatsu Hospital, Osaka
  - Kansai Electric Power Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Osaki Citizen Hospital - Furukawahonami, Ōsaki
  - Saga University Hospital, Saga
  - Kitasato University Hospital, Sagamihara
  - Sanai Hospital - Saitama, Saitama
  - Tokeidai Memorial Hospital, Sapporo
  - Sapporo Medical University Hospital, Sapporo
  - Japan Community Healthcare Organization Hokkaido Hospital, Sapporo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku
  - National Center for Global Health and Medicine, Shinjyuku-ku
  - Tokuyama Central Hospital, Shūnan
  - National Cerebral and Cardiovascular Center, Suita
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi
  - Shizuoka Medical Center, Sunto-gun
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Higashi Takarazuka Satoh Hospital, Takarazuka
  - Takasago Seibu Hospital, Takasago
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Sekino Hospital, Toshimaku
  - Toyama University Hospital, Toyoma
  - Tsuchiura Kyodo General Hospital, Tsuchiura
  - National Hospital Organization Shinshu Ueda Medical Center, Ueda
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama
  - Yokosukakyosai, Yokosuka
- Mexico (42):
  - Centro de Investigación Cardiometabólica de Aguascalientes, Aguascalientes
  - Fundación Cardiovascular de Aguascalientes A.C., Aguascalientes
  - Hospital Cardiologica Aguescalientes, Aguascalientes
  - Enclifar Ensayos Clínicos Farmacológicos Sc, Chihuahua City
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
  - CHRISTUS Centro de Excelencia en Investigación (Norte), General Escobedo
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara
  - Diseno y Planeacion en Investigacion Medica, Guadalajara
  - Centro de Investigacion Medica Integral, Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA S.C., Guadalajara
  - Virgen Cardiovascular Research SC, Guadalajara
  - CINVEC Medica, Guadalajara
  - Investigación Médica Sonora, S.C., Hermosillo
  - Instituto Cardiovascular de León S.C., León
  - RM Pharma Specialists, Mexico City
  - Clínicos Asociados BOCM, Mexico City
  - Grupo Medico Camino Sc, Mexico City
  - Hospital de Jésus, I.A.P., Mexico City
  - Clinica Omega, Mexico City
  - Centro Médico Nacional Siglo XXI, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City
  - ProcliniQ Investigación Clínica SA de CV, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Medical Care and Research SA de CV, Mérida
  - Clinstile, S.A. de C.V., México
  - Accelerium Clinical Research, Monterrey
  - Cardiolink Clin Trials, Monterrey
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
  - UBAM Unidad Biomedica Avanzada Monterrey, Monterrey
  - Clínica García Flores SC, Monterrey
  - Centro de investigación y control metabólico, Monterrey
  - Clinica de Enfermedades Crónicas y de Procedimientos Especiales, Morelia
  - Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro
  - PanAmerican Clinical Research - Querétaro - Avenida Antea, Querétaro
  - Centro de Atención e Investigación Cardiovascular del Potosí, San Luis Potosí City
  - Servicios Integrales Nova de Monterrey S.A. de C.V., San Nicolás de los Garza
  - Centro de Investigacion Cardiovascular y Metabólica, Tijuana
  - Medimanage Research, Tlalpan
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
  - Hospital Angeles Xalapa, Xalapa
- Netherlands (30):
  - Meander Medisch Centrum, Amersfoort
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Rode Kruis Ziekenhuis, Beverwijk
  - Reinier de Graaf Ziekenhuis, locatie Delft, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Admiraal de Ruyter Ziekenhuis, locatie Goes, Goes
  - Groene Hart Ziekenhuis, Gouda
  - General Practitioners Research Institute (GPRI), Groningen
  - Martini Ziekenhuis, Groningen
  - Spaarne Gasthuis, Haarlem Zuid, Haarlem
  - Saxenburgh Medisch Centrum, Hardenberg
  - Ziekenhuis St. Jansdal, Harderwijk
  - Tergooiziekenhuizen, locatie Hilversum, Hilversum
  - Medische Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Radboudumc, Nijmegen
  - Bravis Ziekenhuis, locatie Roosendaal, Roosendaal
  - Erasmus Medisch Centrum, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Antonius Ziekenhuis, locatie D&A Research and Genetics, Sneek
  - Haga Ziekenhuis locatie Leyweg, The Hague
  - ETZ TweeSteden, Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Maxima Medisch Centrum, locatie Veldhoven, Veldhoven
  - VieCuri Medisch Centrum, locatie Venlo, Venlo
  - Zaans Medisch Centrum, Zaandam
- Poland (31):
  - Specderm Poznanska sp.j., Bialystok
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Centrum Medyczne INTERCOR Sp. z o.o., Bydgoszcz
  - Polsko-Amerykańskie Kliniki Serca PAKS Małopolskie Centrum Sercowo-Naczyniowe, Chrzanów
  - Polsko-Amerykańskie Kliniki Serca, Dąbrowa Górnicza
  - Centrum Kliniczno-Badawcze, Elblag
  - NZOZ Twoje Zdrowie EL Sp. z o. o., Elblag
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Przychodnie Grudziądz, Grudziądz
  - NZOZ Salvia CM, Katowice
  - Polsko-Amerykańskie Kliniki Serca, Kędzierzyn-Koźle
  - Centrum Medyczne Linden, Krakow
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - Poliklinika Kardiologiczna Serce, Leszno
  - Centra Medyczne Medyceusz, Lodz
  - Pro Salus Centrum Medyczne, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Clinical Best Solutions, Lublin
  - 1 Wojskowy Szpital Kliniczny w Lublinie, Lublin
  - CenterMed Lublin NZOZ, Lublin
  - Private Practice - Dr. Michał Tomaszewski, Lublin
  - Wielospecjalistyczny Szpital Samodzielny Publiczny Zakład Opieki Zdrowotnej w Nowej Soli, Nowa Sól
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl
  - AKA-MED Centrum, Ruda Śląska
  - Centrum Szybkiej Diagnostyki Kardiologicznej "Kardiomed" M. Żabówka E. Żabówka, Tarnów
  - Polsko-Amerykańskie Kliniki Serca, Tychy
  - Clinical Best Solutions, Warsaw
  - Balsam Medica, Warsaw
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Wroclaw
  - NZOZ Centurm Medyczne SERAFIN-MED, Żarów
- Puerto Rico (2):
  - Advanced Clinical Research, LLC, Bayamón
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
- Romania (23):
  - CMI Cardiologie - Dr. Mercea Corina Delia, Baia Mare
  - CMI DNBM Dr. Pop Lavinia, Baia Mare
  - C.M.D.T.A. Neomed, Brasov
  - Nicodiab, Bucharest
  - Hightech Medical Services SRL-Centrul pentru Studiul Metabolismului, Bucharest
  - Centrul Medical NutriLife, Bucharest
  - Spitalul Universitar de Urgență București, Bucharest
  - Centrul Medical Endocrinologie si Diabet Dr. Paveliu, Bucharest
  - Mat Cord Biomedica S.R.L., Buzău
  - Spitalul Clinic Județean de Urgență, Craiova
  - Milena Sante, Galați
  - Diamed Obesity, Galați
  - Centrul Medical Consultmed, Iași
  - Cardiomed Iași, Iași
  - Clinica Korall, Satu Mare
  - Policlinica Astra Sibiu, Sibiu
  - SC Dentosim Queen SRL - Centrul Medical Diamed, Târgu Mureş
  - Cardiomed, Târgu Mureş
  - Centrul Medical Mediab, Târgu Mureş
  - Mediab S.R.L., Târgu Mureş
  - Private Practice - Dr. Cristian Podoleanu, Târgu Mureş
  - Cabinet Medical Dr.Geru, Timișoara
  - Institutul de Boli Cardiovasculare Timișoara, Timișoara
- Slovakia (14):
  - Cliniq s.r.o., Bratislava
  - ENDIAMED s.r.o, Dolný Kubín
  - JM-Interna s.r.o, Dolný Kubín
  - IN-DIA, Lučenec
  - NEDÚ - Národný endokrinologický a diabetologický ústav n.o., Ľubochňa
  - Sin Azucar, Malacky
  - AMBORA s.r.o. Interna ambulancia, Martin
  - Fakultná nemocnica Nitra, Nitra
  - MEDIKALS, Piešťany
  - MEDISPOL, Prešov
  - ENRIN, s.r.o., Rimavská Sobota
  - Tatratrial s.r.o., Rožňava
  - Areteus s.r.o., Trebišov
  - MediPrax, s.r.o., Trstená
- South Korea (20):
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Eulji University Hospital, Daejeon
  - Boramae Medical Center, Dongjak-gu
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Sejong General Hospital, Sosa-gu
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
- Spain (43):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Fundacion ALcorcon, Alcorcón
  - Hospital Germans Trias i Pujol, Badalona
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital de Denia Marina Salud, Denia
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol
  - Hospital de Cabueñes, Gijón
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen Nieves, Granada
  - Hospital Infanta Elena, Huelva
  - Hospital Universitario de Jaen, Jaén
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Lucus Augusti, Lugo
  - FutureMeds - Madrid, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitari Son Espases, Palma
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Salut Sant Joan de Reus-Baix Camp (Edp), Reus
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Virgen del Camino, Sanlúcar de Barrameda
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí
  - Hospital Universitario Marqués de Valdecilla, Santander
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Hospital Universitario Virgen Macarena, Seville
  - FutureMeds - Sevilla, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Vithas Hospital Sevilla, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Virgen de las Montañas, Villamartín
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (15):
  - Changhua Christian Hospital, Changhua County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - Fu Jen Catholic University Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
  - National Yang Ming Chiao Tung University Hospital, Yilan
- United Kingdom (17):
  - Layton Medical Centre, Blackpool
  - Bristol Royal Infirmary, Bristol
  - Cheadle Community Hospital, Cheadle
  - Panthera Biopartners - North London, Enfield
  - Panthera Biopartners - Glasgow, Glasgow
  - Hull Royal Infirmary, Hull
  - Royal Free Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Panthera Biopartners - Preston, Preston
  - Panthera Biopartners - Manchester, Rochdale
  - Salford Royal Hospital, Salford
  - Panthera Biopartners - Sheffield, Sheffield
  - Lister Hospital, Stevenage
  - Torbay Hospital, Torquay
  - Sunderland Royal Hospital, Tyne and Wear
  - Sandwell General Hospital, West Bromwich
  - Panthera Clinic - York, York

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Byambaa E, Roshanravan B, Berglund L. Lipoprotein(a) and CKD: Insights into New Therapeutic Opportunities. Clin J Am Soc Nephrol. 2025 Dec 2. doi: 10.2215/CJN.0000000968. Online ahead of print. PMID 41329869
- [Derived] Nicholls SJ. Therapeutic lowering of lipoprotein(a): implications for improving outcomes in patients with peripheral arterial disease. Curr Opin Lipidol. 2025 Oct 1;36(5):232-237. doi: 10.1097/MOL.0000000000001002. Epub 2025 Jul 21. PMID 40699211
- [Derived] Nicholls SJ, Nelson AJ, Michael LF. Oral agents for lowering lipoprotein(a). Curr Opin Lipidol. 2024 Dec 1;35(6):275-280. doi: 10.1097/MOL.0000000000000953. Epub 2024 Sep 25. PMID 39329200
- See also: Related Info — https://trials.lilly.com/en-US/trial/465595